IRAS ID: 271897

**Researchers:** 

Participant Identification Number for this trial:



## **CONSENT FORM**

Effect of short-term negative energy balance on systemic biomarkers associated with osteoarthritic symptoms in early knee osteoarthritis patients.

| Ms Rachel Deere | | Tel: 01225 385918 | email: R.Deere@bath.ac.uk |
|---|---|---|---|
| Dr Enhad Chowdhury | | Tel: 01225 385428 | email: E.Chowdhury@bath.ac.uk |
| Professor James Bilzon | | Tel: 01225 383174 | email: J.Bilzon@bath.ac.uk |
| Please initial box | | | |
| 1. I confirm that I have read the information sheet dated 13/10/2021 (version 2.0) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| 3. | I agree that my samples may be stored and used until all analysis for this study is complete. | | |
| 4. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from within the research team at the University of Bath, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | |
| 5. | I understand that damage caused during the equipment loan is covered by the Universities Insurance, however the University and Research team do not accept responsibility for any damage that may arise as a consequence of machine delivery and use (e.g., superficial damage to flooring and walls). Study enrolment will include an assessment of the practicality of delivering and housing the equipment in your home. | | |
| 6. | I understand that the informa other research in the future a | | • • |
| 7. | I agree for my personal details to be kept on file so I can be contact with information about future research. | | |

taking consent

Date

Date

8. I agree to take part in the above study.

Name of Participant

Name of Person

Signature

Signature